CLINICAL TRIAL: NCT03751956
Title: A Study Evaluating the Mass Balance and Biotransformation of [14C]HSK3486 Emulsion Injection in Healthy Chinese Male Adults.
Brief Title: A Study Evaluating the Mass Balance of [14C]HSK3486 Emulsion Injection in Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK3486-104-2
Record Dates: First submitted 2018-11-18; First posted 2018-11-23 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Anesthesia; Sedation
MeSH Terms: interventions — HSK3486

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HSK3486 (Experimental): 0.8 μCi/0.4 mg/kg of [14C]HSK3486 emulsion injection
  Interventions: Drug: HSK3486

INTERVENTIONS:
Drug: HSK3486 — The subjects will receive an intravenous injection of 0.8 μCi/0.4 mg/kg of [14C]HSK3486 emulsion injection (i.e., a subject with the body weight of 60 kg is administered with a radiation dose of 48 μCi).

SUMMARY:
This study is designed to evaluate the mass balance and biotransformation pathways of HSK3486 in healthy Chinese male subjects administered with a single intravenous dose of [14C]HSK3486, so as to characterize the drug's general pharmacokinetics and safety in humans and provide supportive data for reasonable use.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in this study are required to meet all of the following:

  1. Healthy Chinese males aged 18-49 years old (inclusive);
  2. Body weight: body mass index (BMI) between 19-26 kg/m2 (inclusive); weight should be no less than 50 kg; weight difference between the lightest and the heaviest subjects enrolled should be no more than 10 kg;
  3. Vital signs: blood pressure between 90-140/60-90 mmHg; heart rate or pulse between 60-99 beats/min; body temperature (ear temperature) between 35.5-37.1 °C; respiratory rate between 12-24 breaths/min; blood oxygen saturation when inhaling ≥ 96% (inclusive);
  4. Normal major organ function, e.g. routine blood test, blood biochemistry, routine urinalysis, feces and fecal occult blood test, and blood coagulation are all normal, or abnormal with no clinical significance as judged by the investigators;
  5. Subjects who voluntarily sign the informed consent form, able to communicate well with the investigator and complete all trial procedures in accordance with the protocol.

Exclusion Criteria:

* Subjects who meet any of the following will be excluded:

  1. Subjects with clinically significant abnormalities during screening in physical examinations, laboratory tests, 12-lead ECG, chest X-ray or airway evaluation, including airway evaluation of a modified Mallampati score of IV; subjects with positive test result for hepatitis B surface antigen, hepatitis B e antigen, hepatitis C antibody, HIV antibody or syphilis antibody;
  2. Medication history: In receipt of any other investigational drug or participated in any drug or medical device clinical trial within 3 months before screening; or in receipt of propofol, other sedative/narcotic drugs and/or opioid analgesics or compounds containing analgesics within 72 hours prior to screening; or in receipt of any prescription drugs, Chinese herbal medicines, over-the-counter drugs or food supplements (such as vitamins and calcium supplements) other than contraceptives, paracetamol, oral non-steroidal anti-inflammatory drugs, and topical over-the-counter preparations within 2 weeks before screening; subjects can only be enrolled given the condition that the primary investigator (PI) and the sponsor agree that the drug used has no effect on the safety and mass balance results of the trial;
  3. Past and current medical history:

     A Subjects with a history of any severe disease, or concomitant diseases or abnormalities that may affect the test results as judged by the investigator, including but not limited to diseases or abnormalities in the circulatory system, endocrine system, neurological system, digestive system, urinary system, hematologic system, immune system, mental and metabolic aspects; B Subjects who have a past or current history of cardiovascular disease, including: heart failure, ischemic heart disease, long QT syndrome, arrhythmia requiring medication; a family history of Adams-Stokes syndrome or long QT syndrome; QTcF interval ≥ 450 ms (corrected by Fridericia's formula); C Subjects who have a past or current history of respiratory disease, including: obstructive pulmonary disease, asthma, or a history of bronchospasm requiring treatment within 3 months prior to screening; acute respiratory infections within 1 week prior to screening, with significant fever, wheezing, nasal congestion, and coughing.

     D Subjects who have a past or current history of gastrointestinal disease, including: gastroesophageal reflux, hemorrhoids or perianal disease with fecal blood, habitual constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease, etc.; E Subjects who have major surgery within 6 months before screening, or surgical incision not completely healed. Major surgery includes, but is not limited to any surgery that has a significant risk of bleeding, prolonged general anesthesia, incisional biopsy or significant traumatic injury; F Subjects with hyperactive immune response, including: sensitive to excipients of HSK3486 emulsion injections (soybean oil, glycerin, triglyceride, egg lecithin, sodium oleate and sodium hydroxide), history of drug allergies (including anesthetics), or other allergic diseases (such as allergic to any food ingredient or have special dietary requirements and cannot follow a uniform diet);
  4. Alcohol abuse or history of alcohol abuse within 3 months prior to screening, e.g. > 14 units of alcohol consumption per week (1 unit = 360 mL beer or 45 mL liquor with 40% alcohol or 150 mL wine), or positive result for breath alcohol test at screening;
  5. Consumption of more than 5 cigarettes daily within 3 months before screening or habitual use of nicotine-containing products which cannot be withdrawn during the trial; history of respiratory irritation symptoms caused by smoking;
  6. Chronic drug abuse or use of soft drugs (such as marijuana) within 3 months before screening; or use of hard drugs (such as cocaine, amphetamines, phencyclidine) within 1 year before screening; or any signs of chronic benzodiazepines use (such as insomnia, anxiety) or positive urine drug test during screening;
  7. Habitual consumption of grapefruit juice or excessive tea, coffee and/or caffeinated beverages which cannot be withdrawn during the trial;
  8. Engaged in work requiring long-term exposure to radioactive conditions; or significant radioactive exposure within 1 year prior to the trial (≥ 2 chest/ abdominal CT, or ≥ 3 other types of X-ray tests); or those who have participated in radiolabelling testing;
  9. Fertility planner during the trial period and within 1 year after the completion of the trial, or subjects or their spouses who refuse to take strict contraceptive measures (including taking condom, contraceptive sponge, contraceptive gel, diaphragm, intrauterine devices, oral or injectable contraceptives, subcutaneous implants, etc.) during the trial and within 1 year after the completion of the trial;
  10. Subjects who received blood transfusion within 1 month before screening or who had blood loss or blood donation ≥ 200 mL, or subjects who had plasma donation or plasma exchange within 7 days before the trial;
  11. Subject deemed unsuitable by the investigator for any other reason.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Percentage of cumulative drug excretion of [14C]HSK3486 on biological specimens(urine and faeces) accounting for total radiation drug dose | From the start of administration through 168 hours after administration
  Though collecting different periods of biological specimens(urine and faeces) , detecting their respective drug excretion of [14C]HSK3486，calculating the total cumulative excretion amount and relevant proportion of each kind of specimen(urine or faeces)
Maximum Plasma Concentration [Cmax] of total radioactivity and non-radiolabeled HSK3486 respectively | From the start of administration through 168 hours after administration
  Pharmacokinetic Measures
Time to plasma peak concentration[Tmax] of total radioactivity and non-radiolabeled HSK3486 respectively | From the start of administration through 168 hours after administration
  Pharmacokinetic Measures
Clearance half-life[t1/2] of total radioactivity and non-radiolabeled HSK3486 respectively | From the start of administration through 168 hours after administration
  Pharmacokinetic Measures
Area Under the Curve [AUC] of total radioactivity and non-radiolabeled HSK3486 respectively | From the start of administration through 168 hours after administration
  Pharmacokinetic Measures
The metabolite analysis of [14C]HSK3486 in human body | from the start of administration through 168 hours after administration
  Pharmacokinetic Measures

SECONDARY OUTCOMES:
Number of patients with adverse events and serious adverse events | From the time the subject is being screened to the end of the trial( nearly 168h after drug administration)
  Safety Measures
Blood routine test | At the time of subject is being screened and at the end of study( nearly 168h after drug administration)
  Observe the changes of blood routine test during the whole trial
Urine routine test | At the time of subject is being screened and at the end of study( nearly 168h after drug administration)
  Observe the changes of urine routine test during the whole trial
Blood biochemical examination | At the time of subject is being screened and at the end of study( nearly 168h after drug administration)
  Observe the changes of Blood biochemical examination during the whole trial
Blood pressure | From the time the subject is being screened to the end of the trial( nearly 168h after drug administration)
  Observe the changes of blood pressure during the whole trial
Heart rate or pulse | From the time the subject is being screened to the end of the trial( nearly 168h after drug administration)
  Observe the changes of heart rate or pulse during the whole trial
Respiratory rate or blood oxygen saturation | From the time the subject is being screened to the end of the trial( nearly 168h after drug administration)
  Observe the changes of respiratory rate or blood oxygen saturation during the whole trial
Heart rate of electrocardiogram | From the time the subject is being screened to the end of the trial( nearly 168h after drug administration)
  Observe the changes of heart rate of electrocardiogram during the whole trial
RR interval of electrocardiogram | From the time the subject is being screened to the end of the trial( nearly 168h after drug administration)
  Observe the changes of RR interval of electrocardiogram during the whole trial
QT interval of electrocardiogram | From the time the subject is being screened to the end of the trial( nearly 168h after drug administration)
  Observe the changes of QT interval of electrocardiogram during the whole trial
QTcF interval of electrocardiogram | From the time the subject is being screened to the end of the trial( nearly 168h after drug administration)
  Observe the changes of QTcF interval of electrocardiogram during the whole trial
PR interval of electrocardiogram | From the time the subject is being screened to the end of the trial( nearly 168h after drug administration)
  Observe the changes of PR interval of electrocardiogram during the whole trial
QRS interval of electrocardiogram | From the time the subject is being screened to the end of the trial( nearly 168h after drug administration)
  Observe the changes of QRS interval of electrocardiogram during the whole trial

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affilicated Hospital of Soochow University, Suzhou, China

REFERENCES:
- [Derived] Bian Y, Zhang H, Ma S, Jiao Y, Yan P, Liu X, Ma S, Xiong Y, Gu Z, Yu Z, Huang C, Miao L. Mass balance, pharmacokinetics and pharmacodynamics of intravenous HSK3486, a novel anaesthetic, administered to healthy subjects. Br J Clin Pharmacol. 2021 Jan;87(1):93-105. doi: 10.1111/bcp.14363. Epub 2020 Aug 3. PMID 32415708